CLINICAL TRIAL: NCT05102786
Title: A Multi-Site Study to Assess Actual Use of a Heated Tobacco Product With Four Non-Combusted Cigarette Variants in Current Adult Smokers
Brief Title: CSD210904: Study to Assess Actual Use of a Heated Tobacco Product With Four Non-Combusted Cigarette Variants in Current Adult Smokers
Status: Completed | Type: Observational
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CSD210904
Record Dates: First submitted 2021-10-20; First posted 2021-11-02 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Smoking; Tobacco Use; Tobacco Smoking
MeSH Terms: conditions — Smoking; Tobacco Use; Tobacco Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 40007388 — A non-combusted cigarette used with heated tobacco device 20020064
Other: 40007385 — A non-combusted cigarette used with heated tobacco device 20020064
Other: 40007387 — A non-combusted cigarette used with heated tobacco device 20020064
Other: 40007386 — A non-combusted cigarette used with heated tobacco device 20020064

SUMMARY:
This is a multi-site, open-label, 8-week, prospective observational study, conducted at multiple sites geographically dispersed within the U.S. The purpose of this Actual Use Study (AUS) is to investigate how U.S. adult tobacco consumers 21 to 60 years of age, inclusive, who typically smoke on average (≥5 cigarettes/day) on at least 20 out of the past 30 days will use a heated tobacco product comprising a heating device and four non-combusted cigarette variants (HTP Investigational Product [IP]) over a 6-week Actual Use Period (AUP) in their real-life/naturalistic environment and in the context of typical consumer marketing materials.

DETAILED DESCRIPTION:
Adult smokers will be recruited, and candidate subjects who meet study inclusion criteria and none of the exclusion criteria will give verbal consent for further screening. Candidate subjects will be scheduled to attend an in-person Site Enrollment Visit. Subjects will self-report their ad libitum use of the HTP IP as well as use of combustible cigarettes (CCs) and any other tobacco- or nicotine-containing products (TNPs) on a daily basis using an electronic diary (eDiary).

During a 1-week Baseline Assessment Period (BAP), enrolled subjects will record all CC and any other TNP use in the eDiary. At the end of the BAP, subjects will return to the study site for Site Visit 1 (SV1). At this visit, subjects will be provided the HTP IP for the first two weeks of the AUP.

During the subsequent 6-week observational AUP, subjects can choose to use the HTP IP (or not). Subjects will be instructed to record all daily TNP and CC use in the eDiary. They will return to the site every two weeks during the AUP for an in-person interview, to complete questionnaires and for product accountability and resupply. As with SV1, at Site Visit 2 and 3, subjects will be able to select their preferred HTP IP variants (if desired) for use during the subsequent 2-week AUP. Point of sale materials will be present during subject interactions at SVs. After Week 6 of the AUP, there will be a final site visit and week-long Close Out Period.

In addition to collecting information on daily ad libitum use of HTP IP, TNP and CC use, the study will assess subjective measures for each HTP IP, including product use/misuse and intent to use again (at close of study). Information on intention to quit CC use will be collected at enrollment and at study conclusion. A passive surveillance mechanism will be used to collect information on adverse health experiences.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males or females, 21-60 years old, inclusive, verified with government-issued photo ID.
2. Must be a current smoker of factory-made filtered menthol and/or non-menthol cigarettes, has smoked at least 100 cigarettes in their lifetime, and typically smoke on at least 20 days out of the past 30 days.
3. Smokes, on average, ≥ 5 combustible cigarettes per day (CPD) on days when cigarettes are smoked.
4. Must indicate "an intention to use" the HTP IP after a brief review of product information at the Screening and Enrollment Visit (SEV). Subjects will not try the product at the SEV.
5. Available and interested in participating in an 8-week study about the HTP IP.
6. Able and willing to comply with all study requirements, including questionnaires, the eDiary reporting procedures, and provide valid contact information.
7. Able to read, understand, and willing to sign Informed Consent Forms (ICFs) and complete questionnaires written in English.
8. Has not participated in any tobacco-, vapor-, or nicotine-related research within 3 months of screening.

Exclusion Criteria:

1. Self-reports as currently quitting or intending to quit within the next 3 months all tobacco or nicotine product use ("currently" is defined as within (≤) 30 days prior to signing ICF#1). Those who intend to quit CC only can be enrolled.
2. Female subjects who are currently pregnant or breastfeeding or planning to become pregnant or start breastfeeding within the next 6 months based on self-report.
3. Female subjects who self-report they are not using adequate methods to prevent pregnancy.
4. Self-reports "poor" physical health (based on the five-category Population Assessment of Tobacco and Health (PATH) questionnaire): "In general, how would you rate your physical health?" (Response choices: Excellent, Very Good, Good, Fair, Poor).
5. Self-reports "poor" mental health (based on the five-category PATH questionnaire): "In general, how would you rate your mental health?" (Response choices: Excellent, Very Good, Good, Fair, Poor).
6. Employees of tobacco or vapor companies.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study sample will comprise generally healthy, U.S. adult tobacco consumers 21 to 60 years of age, inclusive, who are regular smokers (≥5 cigarettes/day) on at least 20 of 30 days, who are not currently quitting all Tobacco- and/or Nicotine-containing Product (TNP) use, and who have no intention of quitting all TNP use in the next three months (quitting CC use only is allowable). Once enrolled, subjects confirming an intent to quit all TNP use during the AUP will be discontinued. A recruiting target for younger smokers (21-30 years old) of approximately 15% will be established to ensure that they are sufficiently represented among the enrolled subjects.
Sampling Method: Non-Probability Sample
Enrollment: 1180 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Number and Proportion of Established Users | 6 weeks
  Number and proportion of subjects who meet the definition of "established users" of the HTP IP
Number and Proportion of Established Users who reduce their CPD consumption | 8 weeks
  Number and proportion of subjects among "established users" of the HTP IP who reduce their CPD consumption by at least 50%
Descriptive weekly average CPD consumption | 8 weeks
  Descriptive weekly average CPD consumption per subject among all subjects who complete the study, including both established and non-established users of the HTP IP

CONTACTS AND LOCATIONS:
Overall Officials: Mandara Shetty, Study Director — BAT/RAIS
Locations (10):
- United States (10):
  - Schlesinger Atlanta, Atlanta, Georgia
  - Schlesinger Chicago, Chicago, Illinois
  - Schlesinger Baltimore, Baltimore, Maryland
  - Schlesinger Minneapolis, Edina, Minnesota
  - Schlesinger Kansas City, Kansas City, Missouri
  - Schlesinger St. Louis, St Louis, Missouri
  - Schlesinger Charlotte, Charlotte, North Carolina
  - Schlesinger Nashville, Nashville, Tennessee
  - Schlesinger Dallas, Dallas, Texas
  - Schlesinger Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No